CLINICAL TRIAL: NCT06291168
Title: Comparison of The Effectiveness of Chiropractic Manipulation and Yoga-Based Exercise Approach in Patients With Chronic Low Back Pain
Brief Title: Comparison of The Effectiveness of Spinal Manipulation and Yoga in Chronic Low Back Pain
Acronym: CTESMYCLBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Assistant Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CMT002
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain; Spinal Manipulation; Yoga
Keywords: Yoga; Chronic Low Back Pain; Chiropractic Manipulation; Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: The 60 participants will be divided into three groups. These groups will be randomly divided into three groups as chiropractic manipulation group (n=20), yoga-based exercise group (n=20) and conventional exercise group (control group) (n=20). Exercise programs will be performed under the supervision of a physiotherapist. Chiropractic manipulation will be applied to the lumbar region and sacroiliac joint in the side lying position. Data will be analyzed in SPSS 29.0 IBM program. Kruskal-Wallis H test will be used for difference analysis between groups, Kruskal-Wallis H test will be used for comparisons between groups by taking the differences between measurement times and the significance level will be determined as p<0.05.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chiropractic Manipulation (CM) Group (Experimental): Sacroiliac joint manipulation and manipulations to be applied to the lumbar region will be applied twice a week for 8 weeks in the side lying position.
  Interventions: Other: Chiropractic Manipulation (HVLA - High Velocity Low Amplitude)
- Yoga-based Exercise (YBE) Group (Experimental): Yoga treatment includes exercise, respiration, balance and coordination, and stretching and will be performed by a physiotherapist with yoga certification.
  Yoga exercises will be practiced with the classical yoga program, divided into groups of 3-4 people, for 8 weeks, 2 days a week, 60 minutes a day.
  Interventions: Other: Yoga-Based Exercise Program
- Conventional Exercise (Control) Group (CG) (Experimental): Spinal stabilization exercises for the lumbar region will be given in 3 phases following the protocol given to the chiropractic manipulation group. The exercises will be performed two days a week under the supervision of a physiotherapist. Individuals will be called to the hospital two days a week for 8 weeks and will be advised to continue the exercises during the follow-up period. At the end of the 12th week, the exercises will be repeated and progressed with the physiotherapist.
  Interventions: Other: Conventional Exercises

INTERVENTIONS:
Other: Chiropractic Manipulation (HVLA - High Velocity Low Amplitude) — Participants in the groups receiving DNS will be asked to hold the lower leg in the side lying position with the lower leg in the extended position and to clamp the upper leg to the lower leg with hip and knee flexion. During the application, the HLVA technique will be applied once by positioning the hypothenar part of the physiotherapist's hand on the transverse process of the lumbar vertebra where tenderness is felt by palpation and vertebral subluxation is thought to be present.
  After determining that the movement disorder of the sacroiliac joints of the participant is caused by the impaired movement of the ilium in the posterior and inferior direction or the impaired movement of the ilium in the anterior and superior direction, the participant will be asked to take a side lying position.HVLA spinal manipulation was performed for less than one second from posterior to anterior, inferior to superior and medial to lateral directions.
  Arms: Chiropractic Manipulation (CM) Group
Other: Yoga-Based Exercise Program — Yoga treatment includes exercise, respiration, balance and coordination, and stretching and will be performed by a physiotherapist with yoga certification. Patients will be evaluated before treatment, two weeks later, after treatment (at the end of the 8th week) and at the end of the 12th week after treatment (control).
  Yoga exercises will be practiced with the classical yoga program, divided into groups of 3-4 people, for 8 weeks, 2 days a week, 60 minutes a day.
  It will be applied as a yoga session program including breathing and warm-up exercises, suyanamaskar, various relaxation techniques and asanas.
  Arms: Yoga-based Exercise (YBE) Group
Other: Conventional Exercises — Spinal stabilization exercises for the lumbar region will be given in 3 phases following the protocol given to the chiropractic manipulation group. The exercises will be performed two days a week with a physiotherapist. In order to facilitate the memorization and follow-up of the exercises, short videos will be made to facilitate compliance with the exercises by showing the exercises and methods of prevention of low back pain. Individuals will be called to the hospital two days a week for 8 weeks.
  Arms: Conventional Exercise (Control) Group (CG)

SUMMARY:
The aim of our study was to compare the effectiveness of chiropractic manipulation and yoga-based exercise techniques on pain, functionality, depression and anxiety in patients with long-term low back pain.

DETAILED DESCRIPTION:
The study will include 60 individuals between 18 and 65 who meet the inclusion criteria. Demographic and anthropological information will be recorded before starting the study. After these measurements, the participants will be randomly divided into three groups. These groups will be formed as chiropractic manipulation group (n=20), yoga-based exercise group (n=20) and conventional exercise group (control group) (n=20).

In the chiropractic manipulation group, chiropractic manipulation (HVLA maneuver) will be applied to the facet joints of the lumbar vertebrae and the sacroiliac joint 2 times a week for eight weeks.

The yoga-based exercise group will exercise with an exercise program that includes balance, coordination and stretching exercises. Yoga exercises will be done in groups of 3-4 people, including breathing exercises and various relaxation techniques, and will be done in 60-minute sessions 2 days a week for 8 weeks. This will include yoga techniques such as suyanamaskar and asana.

The control group will perform stabilization exercises for the lumbar region. These exercises will be given in 3 phases following the protocol given to the chiropractic manipulation group. The exercises will be explained to the participants via video. Individuals will perform this exercise program 2 days a week for 8 weeks.

Participants will then be assessed using the Numeric Pain Scale, Roland Morris Disability Questionnaire for functional status, Hospital Anxiety and Depression Scale for quality of life and range of motion of the hip and lumbar region.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Experiencing low back pain for at least 3 months
* Pain above 3 on the numeric pain scale
* The patient diagnosed with chronic low back pain by a specialist doctor does not have any contraindications to chiropractic applications
* No contraindications to exercise (systemic diseases, neurological diseases, etc.)
* Patients without joint-related listhesis, spinal stenosis and active discopathy
* Signing the voluntary consent form

Exclusion Criteria:

* Having a fracture or dislocation of the spine,
* Presence of malignancy and infectious disease
* Presence of joint-related listhesis, spinal stenosis and active discopathy
* Presence of osteoporosis
* Those with a history of trauma within at least 3 months
* Pregnancy and suspected pregnancy
* Individuals with inflammatory low back pain
* Those who have undergone surgery and have neurological loss.
* Those with psychiatric problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | It will be used for all groups before starting treatment, at 2 weeks and 8 weeks after starting treatment and at the completion of 12 weeks post-treatment.
  The numeric rating scale is a pain screening tool commonly used to assess current pain intensity using a 0-10 scale, with zero meaning "no pain" and 10 meaning "worst pain imaginable". Numbers from zero to ten are placed on the visual pain scale. It will be used to subjectively measure patients' pain levels.
Roland-Morris Disability Questionnaire | It will be used for all groups before starting treatment, at 2 weeks and 8 weeks after starting treatment and at the completion of 12 weeks post-treatment.
  The Roland Morris Disability Questionnaire consists of 24 items related to low back pain and related perceptions of disability and is a scale used to determine functional status and disability. The questionnaire includes items related to physical ability, activity, home management, eating, psychosocial, sleep/rest and pain frequency. For each item, there are two Yes/No responses. A score of 1 is given for yes and 0 for no. The final score is obtained by summing the scores of the data obtained.
Hospital Anxiety and Depression Scale (HADS) | It will be used for all groups before starting treatment, at 2 weeks and 8 weeks after starting treatment and at the completion of 12 weeks post-treatment.
  The HADS consists of 14 items. Seven of the items measure anxiety and the remaining seven items measure depression. Odd-numbered items measure anxiety and even-numbered items measure depression. The response format provides four response options that are scored on a 0-3 scale. This results in scale values between 0 and 21 for this scale.
Range of Motion (ROM) | It will be used for all groups before starting treatment, at 2 weeks and 8 weeks after starting treatment and at the completion of 12 weeks post-treatment.
  Range of motion is the movement potential of a joint from full extension to full flexion. Measuring the degree of joint mobility is an important guide in the assessment of injury. Range of motion, also known as ROM, is a measure of flexibility involving ligaments, tendons, muscles, bones and joints, so ROM testing plays an essential role in determining fitness and assessing potential damage. Bilateral leg and hip extension and flexion, bilateral hip adduction and abduction, internal and external rotation angles, lumbar extension, flexion and lateral flexion angles of motion will be measured bilaterally.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA HAKTAN HATIK, Study Director — Sinop University